CLINICAL TRIAL: NCT03378986
Title: Functional Recovery After Monolateral or Bilateral Total Hip Arthroplasty
Brief Title: Recovery After Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: CLF17/02
Record Dates: First submitted 2017-12-01; First posted 2017-12-20 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2017-12

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unilateral THA: Patients who underwent to unilateral total hip arthroplasty
  Interventions: Procedure: Unilateral total hip arthroplasty
- Bilateral THA: Patients who underwent to simultaneous bilateral total hip arthroplasty
  Interventions: Procedure: Simultaneous bilateral total hip arthroplasty

INTERVENTIONS:
Procedure: Unilateral total hip arthroplasty — Replacement of one hip joint through a mininvasive surgical procedure
  Groups: Unilateral THA
Procedure: Simultaneous bilateral total hip arthroplasty — Replacement of both hip joints through one-stage mininvasive surgical procedure
  Groups: Bilateral THA

SUMMARY:
This is an observational prospective study aimed to assess the lower limbs motor and functional recovery in patients who underwent to unilateral THA respect to simultaneous bilateral THA, in early postoperative phase.

DETAILED DESCRIPTION:
Introduction: Total hip arthroplasty (THA) represents a successful treatment for several hip joint pathologies. In case of bilateral hip joint involvement, the advancements in surgical techniques have made the development of bilateral THA surgery possible through one-stage procedure. This approach seems to be as safe as unilateral THA and safer than two-stage bilateral THA, but few studies considering functional outcomes in these patients without exploring outcomes linked to their motor and functional performance.

Objective: the aim of the study is to assess the lower limbs motor and functional recovery in patients who underwent to unilateral THA respect to simultaneous bilateral THA, in early postoperative phase.

Methods: 20 patients underwent to unilateral THA and 20 patients underwent to simultaneous bilateral THA will be recruited in the study. The partecipants will be aged from 40 to 65 years old, they will be undergone to primary THA for arthritis and the will be able to walk for 50 m without aids. Patients with severe dysplasia (Crowe III and IV), anchylosis, sub-anchylosis or surgical fusion of the coxophemoral joint, with traumatic event, or previous femoral and / or pelvic osteotomy, will be excluded from the study. Weight distribution and postural stability will be evaluated asking to participants to stay on two stabilometric platform with open eyes and closed eyes for 45 seconds. Gait analysis will be used to evaluate the spatio-temporal gait parametres and the ankle, knee, hip and pelvic kinematic. Pain during walking and patients' walking ability will be also evaluated throught Numeric Rating Scale (NRS) and Timed Up and Go test (TUG). Outcome measures will be collected the day before surgery, after three, seven and about forty days after surgery, except for gait analysis and Time Up and Go tests, which will not be recorded after three days.

Statistical analysis: normality and homogeneity of demographic variables and outcome measures at the baseline will be verified. Intergroup and intra-group post-intervention differences related to outcome measures will be investigated through ANOVA for repeated measurements including post hoc analysis.

ELIGIBILITY:
Inclusion Criteria:

* from 40 to 65 years old
* primary THA for osteoarthritis
* ability to walk for 50 m without aids

Exclusion Criteria:

* severe dysplasia (Crowe III and IV)
* anchylosis, sub-anchylosis or surgical fusion of the coxophemoral joint
* traumatic event
* previous femoral and / or pelvic osteotomy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients who undergone to unilateral THA and 20 patients who undergone to simultaneous bilateral THA
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Weight Distribution | Before surgery, 3rd and 7th postoperative day
  Ability to simmetrically load their lower limbs
Change in Centre of Pressure Length of Trace | Before surgery, 3rd and 7th postoperative day
  Ability to mantain balance

SECONDARY OUTCOMES:
Gait analysis | Before surgery and 7th postoperative day
  Spatio-temporal parametres of the gait and joints kinematic
Change in Numeric Rating Scale | Before surgery, 3rd and 7th postoperative day
  Scale for pain assessment ranging from 0 (absence of pain) to 10 (maximum pain)
Change in Timed Up and Go Test | Before surgeryand 7th postoperative day
  Test for evaluating walking ability

CONTACTS AND LOCATIONS:
Locations (1):
- Roberto Gatti, Rozzano, Milan, Italy

DOCUMENTS (2):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03378986/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03378986/SAP_001.pdf